CLINICAL TRIAL: NCT03161236
Title: Assessing Balance Changes Following an Exercise Program Among Middle-Aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gurinder Bains, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5160196
Record Dates: First submitted 2017-03-15; First posted 2017-05-19 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Balance Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home exercise program (Experimental): • The exercise group will follow a home exercise protocol for eight weeks: that involves standing on one foot, walking, and doing wall squats.
  Interventions: Other: home exercise program
- non exercise group (Active Comparator): • The non-exercise group will continue with their usual life style
  Interventions: Other: non exercise program

INTERVENTIONS:
Other: home exercise program — Subjects in the exercise group will be instructed to follow the intervention protocol for eight weeks. The intervention consists of five exercises: standing on one foot, walking heel to toe, heel walking, side kicks, and wall squats. Each exercise will be repeated three times per week for eight weeks.
  Arms: home exercise program
Other: non exercise program — continue usual lifestyle
  Arms: non exercise group

SUMMARY:
This graduate student research study has two purposes; the first purpose is to examine the criterion validity of the Y Balance Test (YBT) with the Limits of Stability Test (LOS) in healthy middle-aged adults. The second purpose is to examine balance changes using the YBT following a home-based exercise program.

DETAILED DESCRIPTION:
4. "Subjects will be healthy female or male middle-aged adults who are able to walk and move independently.

5. "Subjects will be between 45 and 64 years of age." 6. "In total, subject participation will last approximately eight weeks. Visit 1 (baseline): 90 minutes, visit 2 (week 4): 30 minutes, and visit 3 (week 8): 60 minutes.

7. "Subjects will be recruited by distributing flyers in the Loma Linda Community, sending emails to school staff, students, and faculty, and word of mouth.

8. "Consent will take place at Loma Linda University, Nichol Hall rooms A620 -A640 by investigators." 9. If Multi-center: N/A 10. If Single center or investigator-initiated: "70 subjects will participate in the study."

ELIGIBILITY:
Inclusion Criteria:• Healthy adults.

* Age range: 45-64 years.
* Able to walk and move independently

Exclusion Criteria:• Dizziness, visual or neurological disorders that prevent the ability to complete the testing protocol.

* Lower limb injury in the last 3 months.
* Lower limb surgery in the last 6 months.
* Current involvement in a rehabilitation program.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Y Balance Test | change from baseline to 4 weeks
  The test assesses performance during single-leg balance with a reaching task in the anterior (ANT), posteromedial (PM), and posterolateral (PL) directions to determine lower extremity movement asymmetry and balance deficits. ANT, PM, and PL are a composite measurement.
Y Balance Test | change from 4 weeks to 8 weeks
  The test assesses performance during single-leg balance with a reaching task in the anterior (ANT), posteromedial (PM), and posterolateral (PL) directions to determine lower extremity movement asymmetry and balance deficits. ANT, PM, and PL are a composite measurement.

SECONDARY OUTCOMES:
limits of stability | change from baseline to 4 weeks
  Limits of Stability measure five parameters: reaction time (RT), movement velocity (MVL), endpoint excursion (EPE), maximum excursion (MXE), and directional control (DC). RT, MVL, EPE, MXE, and DC are composite measures.
limits of stability | change from 4 weeks to 8 weeks
  Limits of Stability measure five parameters: reaction time (RT), movement velocity (MVL), endpoint excursion (EPE), maximum excursion (MXE), and directional control (DC). RT, MVL, EPE, MXE, and DC are composite measures.

CONTACTS AND LOCATIONS:
Overall Officials: Gurinder Bains, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No